CLINICAL TRIAL: NCT07223697
Title: An Extension Study To Evaluate the Long-Term Safety and Efficacy of Afimkibart (RO7790121) in Patients With Atopic Dermatitis Who Participated in Previous Afimkibart Clinical Trials
Brief Title: A Long Term Extension Study to Evaluate the Safety and Efficacy of Afimkibart (RO7790121) in Participants With Atopic Dermatitis
Acronym: Velarite-LTE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS45943; 2025-520771-59-00 (EU CTIS Number)
Record Dates: First submitted 2025-10-30; First posted 2025-11-03 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Afimkibart Group I (Experimental): Participants will receive Afimkibart as subcutaneous (SC) injection.
  Interventions: Drug: Afimkibart
- Afimkibart Group II (Experimental): Participants will receive Afimkibart as SC injection.
  Interventions: Drug: Afimkibart

INTERVENTIONS:
Drug: Afimkibart — Afimkibart SC injection will be administered as per the schedule defined in the protocol.
  Other Names: RO7790121; PF-06480605; RVT-3101

SUMMARY:
This study will assess long-term safety and efficacy of Afimkibart (also known as RO7790121) in participants with Atopic Dermatitis (AD) who participated in previous afimkibart clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to comply with all aspects of the protocol including completion of the efficacy assessments (EASI and IGA), clinical outcome assessment instruments (DLQI, POEM), and safety and PK sample collections for the duration of the study

Parent Clinical Trial-Specific Criteria:

* Study CS45570 participants who continued to be evaluated at the Week 36 follow up visit and achieved => EASI50 response from study baseline

Exclusion Criteria:

* Evidence of other skin conditions that would interfere with the assessment of AD
* Withdrawal of consent and/or premature discontinuation from parent study
* Any permanent discontinuation of study drug in parent study
* History of severe allergic reaction or anaphylactic reaction to any biologic agent or known hypersensitivity to any component of Afimkibart

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2033-02-11 (Estimated); Study Completion 2033-02-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events | From Baseline up to 6 years

SECONDARY OUTCOMES:
Change From Baseline (in Parent Study) in Eczema Area and Severity Index (EASI) Score at Each Visit | Baseline, Up to 6 years
Percent Change From Baseline (in Parent Study) in EASI Score at Each Visit | Baseline, Up to 6 years
Percentage of Participants With EASI-50 at Each Visit | Up to 6 years
Percentage of Participants with EASI-75 at Each Visit | Up to 6 years
Percentage of Participants with EASI-90 at Each Visit | Up to 6 years
Percentage of Participants who Achieve Validated Investigator Global Assessment Scale for Atopic Dermatitis (vIGA-AD) of Clear (0) or Almost clear (1) at Each Visit | From Baseline up to 6 years
Change from Baseline (in the parent study) in Participant-Oriented Eczema Measure (POEM) at Each Visit | Baseline, Up to 6 years
Change from Baseline (in the parent study) in Dermatology Life Quality Index (DLQI) at Each Visit | Baseline, Up to 6 years
Serum Concentration of Afimkibart at Specified Timepoints | Pre-dose on Day 1, Weeks 2, 10, 18, 26, 34, 42, 50 74, 98, 122, 146, 170, 194, 218, 242, 266, 290 and 14 weeks after last dose
Percentage of Participants with Anti-Drug Antibodies (ADAs) to Afimkibart | From Baseline up to 6 years
Percentage of Participants with Neutralizing Antibody (NAb) to Afimkibart | From Baseline up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Best Skin Research LLC, Camp Hill, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing